CLINICAL TRIAL: NCT01825343
Title: Preventable Paediatric Trauma - Retrospective Analysis
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Ziv Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: ZIV-0005-13
Record Dates: First submitted 2013-04-02; First posted 2013-04-05 (Estimated); Last update posted 2013-04-05 (Estimated); Status verified 2013-04

CONDITIONS: Pediatric Trauma
Keywords: fall; burn; road traffic crash
MeSH Terms: conditions — Burns

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: None Retained — We are looking retrospectively at data already stored on the hospital database. We have no human subjects and will only analyse hospital records. We will not be contacting patients.
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Purpose: a retrospective study of all Paediatric patients who presented to Ziv Medical Centre with injuries of all systems, major and minor, in order to determine the exact circumstances of the injury, whether this might have been preventable and design a Haddon Matrix of risk factors for injury to target prevention.

Hypothesis: injury prevention interventions can be targetted by finding out local causes of Paediatric Trauma

DETAILED DESCRIPTION:
A Trauma Registry is already kept in the hospital. It is confidential and data is supplied to the government from this registry.

The procedure is to be granted access to the database and access data stored on the mechanism and outcome of Paeditric Trauma. This data will be stored on the work computer of the principal investigator and will be password protected.

Methods: Identify from the Trauma database all patients assessed at Ziv Medical Centre with Trauma, consult their medical notes and document the exact injury, the mechanism of injury, the circumstances, whether the child was alone or supervised, the nature and complications of the injury, treatment required and short and long term progress and disability.

ELIGIBILITY:
Inclusion Criteria:

* All patients classified as Paediatric according to Israeli law (up to the age of 18 years). This includes pregnant women and patients presenting with multiple complaints as well as Trauma, isolated injuries and polytrauma.

Exclusion Criteria:

* Patients for whom no history is available.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Identify from the Trauma database all patients assessed at Ziv Medical Centre with Trauma, consult their medical notes and document the exact injury, the mechanism of injury, the circumstances, whether the child was alone or supervised, the nature and complications of the injury, treatment required and short and long term progress and disability.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2013-04; Primary Completion 2014-04 (Estimated); Study Completion 2014-04 (Estimated)

PRIMARY OUTCOMES:
Establishing exact mechanism of injury | 5 years (2007-2012)
  This is a retrospective study. We approximate that since the Trauma registry began in 2007, there have been 200 Paediatric injuries every year. By the end of this year's data collection, therefore, we estimate that we would have collected data from 1000 patients.

CONTACTS AND LOCATIONS:
Overall Officials: Wajdi Safadi, MD, Study Chair — Specialist Surgeon; Seema Biswas, FRCS, Study Director — Specialist Surgeon; Amram Hadary, MD, Principal Investigator — Senior Surgeon; Igor Waksman, MD, Study Chair — Head of Department; Dudu Fuchs, RN, Study Chair — Ziv Hospital Trauma Coordinator
Locations (1):
- Ziv Hospital, Safed, Galilee, Israel